CLINICAL TRIAL: NCT03870126
Title: Effects of Two Doses of a Plant Extract on Mental and Physical Fatigue
Brief Title: Dose Effect of a Plant Extract on Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-1807
Record Dates: First submitted 2019-02-26; First posted 2019-03-11 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Mental Energy; Physical Performance
Keywords: cognitive; phytochemicals; caffeine; polyphenol; beverage; exercise; mental performance; physical performance; vigilance; vigor; energy; vitality; fatigue; sports performance; high-intensity intermittent exercise
MeSH Terms: conditions — Motor Activity; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Flavored Beverage Mix 1 (Placebo Comparator): Flavored still beverage
  Interventions: Other: Flavored beverage
- Flavored Beverage Mix 2 (Experimental): Flavored still beverage with polyphenols, concentration 1
  Interventions: Other: Flavored beverage
- Flavored Beverage Mix 3 (Experimental): Flavored still beverage with polyphenols, concentration 2
  Interventions: Other: Flavored beverage
- Flavored Beverage Mix 4 (Experimental): Flavored still beverage with caffeine
  Interventions: Other: Flavored beverage

INTERVENTIONS:
Other: Flavored beverage — Consume one beverage at the beginning of each visit of the cross-over sequence

SUMMARY:
Test the short-term effects of the acute consumption of two separate beverages containing different concentrations of polyphenols, a beverage containing 75 mg of caffeine and a flavored placebo beverage on mental energy and physical performance

ELIGIBILITY:
Inclusion Criteria:

* 18-49 years of age
* Self-report of good health
* Physical activity requirement: Recreationally active (exercise ≥3 times per week for >30 minutes per session; both cyclists and non-cyclists may enroll)

Exclusion Criteria:

* Under the care of a physician
* Visual impairment that cannot be corrected with glasses or contact lenses
* Inability to perform high intensity exercise (defined perceptually as exercise that feels at least "hard" and this is usually quantified using the Borg 6 to 20 scale. High intensity cycling exercise is defined objectively as exercise causing a high heart rate, defined as a heart rate that is equal to or greater than 70% of heart rate reserve.)
* Inability to adequately perform the cognitive tasks (i.e., cannot complete the task due to -inability to understand instructions or >50% incorrect responses)
* Presence of current or chronic gastrointestinal, sleep or psychiatric disorder
* Pregnant/lactating
* Current smoker
* Report illegal drug use
* Report hypersensitivity to caffeine
* Food allergies/intolerances/sensitivities (including coffee or related foods/beverages/products)
* Current use of dietary supplements, or prescription medication except for oral contraceptives
* Unwillingness to abstain from over the counter medications (e.g. NSAIDS, allergy medications) and caffeine/coffee/foods high in polyphenols for 12 hours prior to the study
* Unwilling to refrain from consuming apple and grapefruit products on study days and 12 hours prior to test days.
* Participation in another clinical trial within the past 30 days or participation in another PepsiCo trial in the past 6 months

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Subjective mental energy: Cognitive test battery | Baseline and 60 min post treatment
  Changes in subjective measures of mental alertness and mental fatigue through computer administered cognitive test battery domains of short-term memory, attention and mood. Tasks are word presentation, word recognition, picture presentation, picture recognition, Cognitive Demand Battery (CDB) serial 3 and serial 7 subtraction, and Bakan task/Rapid Visual Information Processing (RVIP). Performance measures: % correct, % errors and response time in milliseconds.
Subjective mental energy: VAS for mental alertness | Baseline and 60 min post treatment
  Changes in subjective ratings of mental alertness following computer administered cognitively fatiguing tasks. Visual Analog Scale (VAS) for mental alertness has the score range 0-100 (from not at all to extremely).
Subjective mental energy: VAS for motivation | Baseline and 60 min post treatment
  Changes in subjective ratings of motivation following computer administered cognitively fatiguing tasks. Visual Analog Scale (VAS) for motivation has the score range 0-100 (from not at all to extremely).
Subjective mental energy: VAS for mental fatigue | Baseline and 60 min post treatment
  Changes in subjective ratings of fatigue following computer administered cognitively fatiguing tasks. Visual Analog Scale (VAS) for fatigue has the score range 0-100 (from not at all to extremely).
Subjective mental and physical energy: VAS for mental and physical state and trait energy and fatigue (EFS State Scales) | Baseline and 60 min post treatment
  Changes in subjective ratings of mental alertness, motivation and fatigue following computer administered cognitively fatiguing tasks. Mental and Physical State and Trait Energy and Fatigue Scales (EFS State Scales) consist of 12 VAS items to measure intensity of current feeling of physical energy and fatigue and mental energy and fatigue (3 sub-scales each). Score range: The 3 items from each sub-scale are summed and scores for each sub-scale range from 0-300 (none to strongest).
Subjective mental energy: VAS for mood | Baseline and 60 min post treatment
  Changes in subjective ratings of mental alertness, motivation and fatigue following computer administered cognitively fatiguing tasks. The Bond-Lader test uses 16 Visual Analog Scales (VAS) to measure different aspects of mood, with score range 0-100 for each scale (from absence of feeling to presence of feeling).
Subjective mental energy: VAS for caffeine symptoms | Baseline and 60 min post treatment
  Changes in subjective ratings of mental alertness, motivation and fatigue following computer administered cognitively fatiguing tasks. Caffeine symptoms are measured on paper using 8 Visual Analog Scales (VAS) with score range 0-100 (from not at all to extremely).

SECONDARY OUTCOMES:
Physical performance | During the last 3 minutes of 23 min high intensity cycling exercise (10 x 1 min work intervals each followed by 1 min rest. No rest after final interval, 3 min max power from minutes 20-23.
  Mean power output in a timed cycling trial following post-treatment cognitive test battery and caffeine symptom VAS.
Physical Fatigue | After each of 10 1-minute high intensity cycling intervals separated by 1 min rest and at end of exercise.
  Subjective categorical scale, score range 0-7, higher score indicates greater feeling of physical fatigue
Alertness | After each of 10 1-minute high intensity cycling intervals separated by 1 min rest and at end of exercise.
  Subjective categorical scale, score range 1-7, higher score indicates greater alertness meaning a greater feeling of energy
Effort | After each of 10 1-minute high intensity cycling intervals separated by 1 min rest and at end of exercise.
  Subjective categorical scale, Borg Ratings of Perceived Exertion (RPE) measures perception of effort, score range 6-20. Higher score indicates greater effort. 17 or greater generally indicates maximal effort
Quadriceps muscle pain | After each of 10 1-minute high intensity cycling intervals separated by 1 min rest and at end of exercise.
  Subjective categorical scale with ratio-like properties, scale 0-10 with open-ended option for ratings greater than but proportional to 10. Higher scores indicate greater perception of pain in the quadriceps

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J O'Connor, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be kept securely at U. Georgia for several years and can be accessed upon request by contacting Dr. Pat O'Connor (poconnor@uga.edu)
Time Frame: After publication
Access Criteria: Open access, upon request